CLINICAL TRIAL: NCT05008627
Title: PERSONAL PROTECTION EQUIPMENT AND SARS-CoV-2 CONTAMINATION: An Observational Quality Control Study
Brief Title: PERSONAL PROTECTION EQUIPMENT AND SARS-CoV-2 CONTAMINATION
Status: Completed | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, LUIS GAITINI MD, Associate Clinical Professor of Anesthesiology, Bnai Zion Medical Center
Other Study IDs: 0059-21-BNZ
Record Dates: First submitted 2021-08-15; First posted 2021-08-17 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Contaminated Medical or Biological Substances
Keywords: VIRAL CONTAMINATION; DOFFING PPE; GUIDELINES FOR DOFFING

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Doffing PPE with verbal instructions and monitor: The subject will remove the PPE according to verbal instructions by a monitor
- Doffing PPE without verbal instructions: The subject will remove the PPE independently without a monitor

SUMMARY:
Transmission of SARS-CoV-2 occurs through common routes, aerosols and medical procedure.

Personal protective equipment (PPE) reduces the risk of contamination. The risk of contamination of skin and clothing may be particularly high during removal PPE.

The Ministry of Health (MOH) of Israel adapted the technique of using a supervisor that monitors during removal of the PPE.

The aim of this study to examine the using the pre-established protocol, where a staff member removing the PPE according supervision by a staff monitor in comparison with removing the PPE without being instructed neither supervised.

The Protocol provided by MOH is in accordance with the recommendations of the Centers for Disease Control United States (CDC), was presented to all staff.

Study population will include 49 participants: 7 nurses, 7 clinician physicians, 7 cleaning personal, 7 X-rays technicians, 7 anesthesia technician and 7 physiotherapists 7 stretcher bearers, will performed this quality control observational study.

The trail processes of doffing the PPE will be performed twice, first in the present of a trained supervisor and verbal instructions and once again independently in the absence of supervision.

After donning the routine uniform with a new PPE, then the subject will be asked to transfer to an area were the participant's' PPE will be "contaminated" (in the same areas in all participants: over the thorax, shoulders, arms, hands legs and Face Shield) using a brush tool, with the 'Glo' Germ Solution that simulates contamination with a virus on the PPE. The 'Glo' Germ Solution is a non toxic, odorless gel, which glows brightly in the dark when exposed to ultraviolet light to simulate contamination with the virus.

To proceed, the participant will be asked to move a step aside to another area. There the participant will remove the PPE.

After the removal of the PPE the participant will be examined in a dark plot in order to detect a probably contamination traces with the 'Glo' Germ solution that will be illuminated under the ultraviolet UV light.

The participant will repeat the procedure from the beginning, following all stages only in this second time without following the supervisor verbal instructions.

In both trails, after the PPE removal, Ultraviolet Lamp will be used in order to check if the participant had been contaminated in any part of the body or cloth with the 'Glo' Germ Solution

DETAILED DESCRIPTION:
PERSONAL PROTECTION EQUIPMENT AND SARS-CoV-2 CONTAMINATION: An observational quality control study Human-to-human transmission of SARS-CoV-2 (COVID-19) occurs through common routes such as direct transmission, contact transmission and airborne transmissions as aerosols and during medical procedure.

Personal protective equipment (PPE) reduces, but does not eliminate, the risk of skin and clothing contamination with a virus among health care personnel. High-risk exposures, such as prolonged exposure, handling contaminated body fluids, and failure to correctly use PPE, increases the risk of contamination.

The risk of inadvertent contamination of skin and clothing may be particularly high during removal of contaminated PPE.

It was presented that during PPE removal, the subject, especially the dorsum of his hands, were contaminated and virus was transferred to the palms hands and clothing.

Operating protocols recommended by the Centers for Disease Control and Prevention (CDC) have been associated with less frequent hand and clothing contamination compared with no standardized methods, suggesting that the use of the appropriate technique can reduce contamination. Another potential measure to reduce contamination during PPE removal is in the present of a trained supervisor monitoring each step of the removal process, as has been recommended when caring for patients with suspected or confirmed Ebola virus infection.

The Ministry of Health (MOH) of Israel adapted the technique of using a supervisor to guide the medical personal that work in the Covid Unit during donning and doffing the PPE.

A quality controlled observational study will be performed to examine if using visual vigilance control and verbal oral instructions to remove the contaminated PPE, in an appropriate technique, that prevents or reduces contamination during the procedure, in comparison with performing the removal of the PPE independently without visual control and verbal instructions by in the absence of supervisor.

The aim of this study to examine the using the pre-established protocol, where a staff member removing the PPE according to the visual supervision by a staff monitor and follows the instructions carefully, in comparison with the removing the PPE without being instructed neither supervised.

The study received the approval of the Bnai-Zion Medical Center, Haifa, Israel, Ethic Committee No 0059-21-BNZ.

Statistical Analysis A 1% of contamination will be considered as an acceptable level and 10% of contamination as a non-acceptable level. To detect such deviation from the acceptable level in a Z-test on the proportion of contamination with 95% power and one-sided α of 0.05, 34 participants be required.

Materials and Methods Before opening of the Corona Unit at the Hospital, the Infected Disease Department provided educational sessions for personnel from long term care facility. The session included 15 minutes video presentation and practicing of PPE donning and doffing technique.

The protocol provided by the MOH according with CDC recommendations was presented to all staff. A poster highlighting the instructions was displayed throughout the Corona Unit. Based on national recommendations, a checklist including 10 instructions (See Appendix 1) were compiled, it contained items to assess the processes of doffing of the PPE with the necessary work steps such as the required of hand disinfection. The Protocol includes additional measures to reduce contamination, during PPE removal. A trained supervisor was observing and giving verbal indication of each step of the removal process. This strategy was used during Ebola epidemic.

The present simulation study will be conducted in the Simulation Unit of the Anesthesiology Department in Bnai Zion Medical Center, Haifa, Israel.

Study population will include 49 participants: 7 nurses, 7 clinician physicians, 7 cleaning personal, 7 X-rays technicians, 7 anesthesia technician and 7 physiotherapists 7 stretcher bearers will performed this quality control observational study.

The trail processes of donning the PPE will be performed twice, first with the present of a trained supervisor and verbal instructions and once again independently in the absence of supervision.

The experiment will be conducted in 3 areas, namely, area A (clean zone), area B (preparation zone), and area C (test zone).

Area A, a clean zone where subjects will donn their clean isolation gown or apron by themselves.

After putting on over the routine uniform a new PPE (Cobes Industries Co Ltd, Hefei, China) gown or apron, NP95 Mask and a face shield, the subject then will be asked to transfer to area B, there participant's' PPE will be "contaminated" in the same areas in all participants: over the thorax, shoulders, arms, hands legs and Face Shield using a brush tool, with the Glo Germ Solution (Glo Germ Lotion, Glo Germ, Moab, Utah, USA) that simulates contamination with a virus on the PPE. The Glo Germ Solution is a non toxic, odorless gel, which glows brightly in the dark when exposed to ultraviolet light to simulate contamination with the virus, including transfer to skin, clothing, and environmental surfaces during PPE removal. (www.amazon.com/Glo Germ-Powder solution).

To proceed, the participant will be asked to move a step aside to area C. There the participant will remove the PPE, boats, the apron, mask NP95 and face shield according the pre-established Protocol under an oral indications by the research staff following the 10 guidance instructions.

The contaminated PPE equipment will be discarded in a dumpster. After the removal of the PPE the participant will be examined in a dark plot in order to detect a probably contamination traces with the Glo Germ solution that will be illuminated under the ultraviolet UV light.

The participant will repeat the procedure, following all stages only in the second time without the following the supervisor verbal instructions.

In both trails, after the PPE removal, Ultraviolet Lamp will be used in order to check if the participant had been contaminated in any part of the body or cloth with the Glo Germ Solution.

All the procedures will be recorded with a I-Phone 8 camera during all the time of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age limit
* Staff members who worked in CORONA UNIT

Exclusion Criteria:

* Staff members who did not work in CORONA UNIT

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Staff members of the CORONA UNIT
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Contamination with simulated virus | 15 minutes
  Quality control observation

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Somri, MD, Study Director — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel